CLINICAL TRIAL: NCT03863704
Title: Transcutaneous Vagal Nerve Stimulation to Treat Pediatric Inflammatory Bowel Disease
Brief Title: Transcutaneous VNS to Treat Pediatric IBD
Acronym: STIMIBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-0945
Record Dates: First submitted 2019-02-14; First posted 2019-03-05 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects will be given two possible anatomic sites to apply nerve stimulation, one of which is known to induce vagal nerve stimulation and the other does not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- nerve stimulation ear then leg (Sham Comparator): Subjects in this arm will be randomized to receive nerve stimulation with TENS of the ear followed by leg stimulation
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- nerve stimulation leg then ear (Sham Comparator): Subjects in this arm will be randomized to receive leg nerve stimulation with TENS followed by ear nerve stimulation
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Subjects receiving Infliximab (Other): Subjects on Infliximab as part of their clinical care will not be randomized as the study treatment for these subjects will be the same. The sham arm is not included for patients on infliximab.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — To apply transcutaneous electrical stimulation using a TENS unit to the ear or the leg.

SUMMARY:
The current available therapies for inflammatory bowel disease (IBD), including immunomodulator and biologic medications may have toxicities limiting use or inadequate effect. We propose a novel approach to the treatment of IBD by using transcutaneous vagal nerve stimulation (VNS). Research has previously identified that VNS using a surgically implanted stimulator can improve symptoms and decrease inflammation in people with inflammatory diseases. This study will evaluate the use of non-invasive nerve stimulation through the skin (rather than through an implanted device) as a potential therapy in pediatric patients with Crohn Disease or ulcerative colitis. We will be evaluating how this nerve stimulation affects symptoms, markers of inflammation found in the blood and stool including cytokine levels, and heart rate variability. The primary hypothesis of the study is the use of transcutaneous VNS will decrease inflammation in people with IBD leading to improved signs and symptoms of disease. The primary endpoint of the study is to evaluate the change in fecal calprotectin after 16 weeks of nerve stimulation. Secondary endpoints include changes in symptom scores, blood cytokine levels, and heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

1. Age 10-21 years
2. IBD diagnosis for at least 3 months, confirmed by clinical, biochemical, and endoscopic evaluations
3. Elevated Fecal calprotectin ≥ 200 ug/g within the past 4 weeks prior to enrollment
4. Evidence of active inflammatory disease despite treatment with at least one conventional therapy
5. If on corticosteroids, the dose must be stable and ≤ 10mg/day (prednisone or equivalent) for at least 14 days before entry into study
6. If on 5-Aminosalicylate, dose must be stable with following parameters:

   * 28 days on oral medication
   * Prior to baseline calprotectin, 28 days on rectal medication or 2 weeks off rectal medication
7. If on background immunosuppressive treatment the dose must be stable with the following parameters:

   * 56 days (8 weeks) for Immunomodulators (methotrexate, 6-MP, Azathioprine)
   * 112 days (16 weeks) for Infliximab, Adalimumab, Vedolizumab, Ustekinumab, other biologic
8. Able and willing to give written informed consent and comply with the requirements of the study protocol.

Exclusion Criteria:

1. Expectation to increase corticosteroids and/or immunosuppressive treatment
2. Presence of bowel stricture with prestenotic dilatation
3. Presence of intra-abdominal or perirectal abscess
4. Pediatric UC activity Index (PUCAI) score ≥ 65 (severe)
5. weighted Pediatric Crohn Disease Activity Index (wPCDAI) score > 57.5 (severe)
6. Active treatment with antibiotics
7. Presence of active intestinal infection or documented infection by stool PCR or culture analysis in the previous 6 weeks
8. Continuous treatment with an anti-cholinergic medication, including over the counter medications
9. Implantable electronic devices such as pacemakers, defibrillators, hearing aids, cochlear implants or deep brain stimulators.
10. Current tobacco or nicotine user (to limit potential confounding effects of exposure to nicotine)
11. Bowel resection surgery within past 90 days prior to study enrollment and on no conventional IBD therapy, or planned surgery within the course of the study
12. Any planned surgical procedure requiring general anesthesia within the course of the study
13. Participation in any other Investigational drug and/or treatment currently or planned during the length of the study
14. Any condition which, in the opinion of the investigator, would jeopardize the subject's safety following exposure to a study intervention
15. Pregnancy or Lactation
16. Comorbid disease with high likelihood of requiring corticosteroid use
17. Inability to comply with study and follow-up procedures
18. Non-English speaking
19. Known cardiac condition causing or with potential to cause arrhythmia

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Fecal Calprotectin | 16 weeks
  Change in fecal calprotectin over time

SECONDARY OUTCOMES:
Change in Whole blood stimulated cytokine levels over time | 16 weeks
  Blood will be collected into 2 tubes, one with no stimulant and the other with lipopolysaccharide (LPS) to stimulate macrophages to produce cytokines. Cytokine levels within the blood will be assessed and compared to baseline levels. The cytokines being assayed include tumor necrosis factor-alpha, Interferon-gamma, Transforming Growth Factor-beta and Interleukins (IL) - 1, 6, 10, 12, 17, 18, 23. Samples will be collected for this analysis at week 0, 2, 4, and 24
Patient Reported Outcome (PRO) | 16 weeks
  PROMIS Pediatric Profile v2.0-25 and PROMIS Parent Proxy v2.0- 25 questionnaires to evaluate the effect of VNS on abdominal pain intensity and interference in daily activities, fatigue, anxiety, depression, physical function and peer relationships
Pediatric Ulcerative colitis activity index (PUCAI) | 16 weeks
  Change in Pediatric ulcerative colitis activity index over time
Weighted Pediatric Crohn Disease activity index (wPCDAI) | 16 weeks
  Change in weighted Pediatric Crohn Disease activity index over time
Physician Global Assessment (PGA) Score | 16 weeks
  Change in physician global assessment score over time
Heart Rate Variability (HRV) | 16 weeks
  Evaluating change in HRV from baseline until study completion

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Sahn, MD, Principal Investigator — Steven & Alexandra Cohen Children's Medical Center - Northwell Health
Locations (1):
- Steven & Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sahn B, Pascuma K, Kohn N, Tracey KJ, Markowitz JF. Transcutaneous auricular vagus nerve stimulation attenuates inflammatory bowel disease in children: a proof-of-concept clinical trial. Bioelectron Med. 2023 Oct 18;9(1):23. doi: 10.1186/s42234-023-00124-3. PMID 37849000